CLINICAL TRIAL: NCT06877416
Title: A Multi-center, Retrospective, Study on Exploring Optimized Sequential Treatment Strategies of Antibody-Drug Conjugates (ADCs) in HER2-Low-Expressing Breast Cancer
Brief Title: Analysis of Exploring Optimized Sequential Treatment Strategies of Antibody-Drug Conjugates (ADCs) in HER2-Low-Expressing Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yalan Yang, Clinical Investigator, Sun Yat-sen University
Other Study IDs: 20252696
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Antibody-drug Conjugates; HER2-low Breast Cancer; Breast Neoplasms
Keywords: Antibody-drug conjugates; HER2-low Breast Cancer; Retrospective Studies
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (8):
- First-line Trastuzumab Deruxtecan → Second-line Sacituzumab Govitecan
  Interventions: Other: Non-intervention research
- First-line Sacituzumab Govitecan → Second-line Trastuzumab Deruxtecan
  Interventions: Other: Non-intervention research
- First-line RC48 → Second-line Trastuzumab Deruxtecan
  Interventions: Other: Non-intervention research
- First-line Trastuzumab Deruxtecan → Second-line RC48
  Interventions: Other: Non-intervention research
- First-line SKB264 → Second-line Trastuzumab Deruxtecan
  Interventions: Other: Non-intervention research
- First-line Trastuzumab Emtansine → Second-line TQB2102
  Interventions: Other: Non-intervention research
- First-line TQB2102 → Second-line Trastuzumab Deruxtecan
  Interventions: Other: Non-intervention research
- First-line RC48 → Second-line TQB2102
  Interventions: Other: Non-intervention research

INTERVENTIONS:
Other: Non-intervention research — Non-intervention research

SUMMARY:
This study retrospectively analyzes the clinical data of HER2-low breast cancer (IHC 1+/2+ and FISH-negative) patients treated with sequential antibody-drug conjugates (ADCs). Key variables include patient demographics, tumor characteristics, ADC regimens (e.g., trastuzumab deruxtecan, sacituzumab govitecan), treatment sequencing, survival outcomes, and safety profiles. Genomic data (e.g., HER2 expression dynamics, TROP2 levels) are integrated to explore resistance mechanisms and prognostic biomarkers.mechanisms.

This study aims to investigate the efficacy of different ADC sequential regimens in HER2-low breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is one of the most common malignancies in women, posing a significant threat to female health. According to current molecular subtypes, breast cancer is classified into hormone receptor-positive, HER2-positive, and triple-negative breast cancer. However, with the development of novel therapeutic strategies such as antibody-drug conjugates (ADCs), increasing attention has been directed toward HER2-low breast cancer (defined as HER2 immunohistochemistry [IHC] 1+ or 2+/FISH-negative), which accounts for approximately 60%-70% of breast cancer cases. ADCs can exert potential therapeutic effects in HER2-low breast cancer through the "bystander effect" and have been widely adopted in clinical practice. Nevertheless, the optimal sequential treatment strategy for HER2-low patients remains unclear, with a lack of definitive clinical guidelines and limited understanding of resistance mechanisms.

This study aims to investigate the efficacy of different ADC sequential regimens in HER2-low breast cancer patients and explore potential resistance mechanisms. By conducting a retrospective analysis of clinical data from HER2-low patients treated with sequential ADCs, the investigators will evaluate the therapeutic outcomes and safety profiles of various ADC sequencing approaches. Additionally, integrating genomic profiling with routine clinical data, the investigators seek to identify prognostic biomarkers and elucidate resistance pathways. The findings are expected to guide personalized treatment strategies for HER2-low breast cancer patients, ultimately improving clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HER2-low breast cancer, defined as immunohistochemistry (IHC) score of 1+ or IHC score of 2+ with negative in situ hybridization (FISH-negative)
* Received sequential administration of two or more ADCs
* Complete data for patient's character, laboratory and imaging test, treatment and follow-up are available.

Exclusion Criteria:

* Concomitant with other tumor components at the time of diagnosis;
* Have a history of any other malignant tumors;
* Lack of complete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with HER2-low breast cancer, defined as immunohistochemistry (IHC) score of 1+ or IHC score of 2+ with negative in situ hybridization (FISH-negative) who received sequential administration of two or more antibody-drug conjugates (ADCs).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of diagnosis until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 24 months.
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen University Cancer, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No